CLINICAL TRIAL: NCT00540878
Title: An Open-Label, Randomized, Five Period Crossover Study to Estimate the Relative Bioavailability of Five Formulations of 400mg SB-751689 (a Calcium-Sensing Receptor Antagonist) Administered as a Single Oral Dose to Healthy Postmenopausal Females
Brief Title: A Study to Estimate the Effect of Formulation on the Relative Absorption of SB-751689 Administered to Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR9108307
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Osteoporosis
Keywords: Formulation Drug Study
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: SB-751689 oral tablets (400 mg)

SUMMARY:
This study will examine the effects of formulation on the relative bioavailability of SB-751689 (400 mg) administered to healthy postmenopausal women. Subjects will receive a single oral dose of each formulation, with five formulations of SB-751689 tested in total. Blood samples will be taken up to 24 hours postdose after each dose administration. This study will provide information for future possible formulation development of SB-751689 for Phase III.

ELIGIBILITY:
Inclusion criteria:

* Healthy postmenopausal women; 40 and 65 years of age, inclusive
* Non-smokers (as defined in exclusion criteria 6 below)
* Body weight > or = 50 kg and BMI within the range 19-32 kg/m2
* Capable of giving written informed consent and complying with the requirements and restrictions listed in the consent form

Exclusion criteria:

* Any clinically relevant biological or physical abnormality found or reported at screening which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study
* A QTc interval of > 450 msec at screening
* Positive urine drug screen at screening
* Positive urine test for alcohol at pre-dose
* Positive for HIV or hepatitis B or C virus at screening
* Urinary cotinine levels indicative of smoking at screening
* History of smoking or use of nicotine containing products within one year of the study or >10 pack-year history of smoking overall
* History of regular alcohol consumption exceeding 7 units/week (1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening
* History of drug abuse within 6 months of the study
* Participation in a clinical study and received a drug or a new chemical entity with 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of the current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs
* Consumption of red wine, grapefruit, grapefruit juice or grapefruit containing products within 14 days prior to the first dose of study medication
* Donation of blood in excess of 500 mL within 56 days prior to dosing
* Evidence of renal, hepatic or biliary impairment
* History of serious gastrointestinal disease
* History of sensitivity to any of the study medications or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of clinically significant cardiovascular disease
* Medical conditions that might alter bone metabolism
* Serum parathyroid hormone (iPTH) test levels outside the reference range at screening
* Liver function tests, parathyroid hormone test or CPK outside the reference range at screening

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-04

PRIMARY OUTCOMES:
AUC and CMAX after a single dose. | after a single dose

SECONDARY OUTCOMES:
Safety and tolerability after single dose. | after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Port Orange, Florida, United States